CLINICAL TRIAL: NCT02220751
Title: Diagnostic Biomarkers Related to Periodontal Disease Activity in Diabetic
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Priscila Paganini Costa, PhD, University of Sao Paulo
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2008/11033-9; 2008/11033-9 (Other Grant/Funding Number: FAPESP2008/11033-9)
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Periodontitis; Type 2 Diabetes Mellitus
Keywords: Periodontal Attachment Loss; Genes; Saliva; Diagnosis
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus, Type 2; Periodontal Attachment Loss; Disease | interventions — Tooth Exfoliation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- chronic periodontitis (Placebo Comparator): Non-surgical periodontal therapy.
  Interventions: Procedure: Non-surgical periodontal therapy
- Chronic periodontitis + type 2 diabetes (Active Comparator): Non-surgical periodontal therapy + systemic doxycycline non-surgical periodontal therapy was associated with systemic doxycycline 100 mg/day, for two weeks after an initial dose of 200 mg, started on the day before first scaling and root planning session.
  Interventions: Drug: non-surgical periodontal therapy + systemic doxycycline
- Control (No Intervention): Periodontal- and systemically healthy patients were included as control group.

INTERVENTIONS:
Drug: non-surgical periodontal therapy + systemic doxycycline — A program of plaque control with dental prophylaxis and oral hygiene instruction, and the scaling and root planning sessions were included in the non-surgical periodontal therapy. The scaling and root planning was performed by the same operator using curettes and an ultrasonic device, and it was inspected for a second operator. Oral hygiene was reviewed after a week and after a month of periodontal disinfection, followed by dental prophylaxis.
  Non-surgical periodontal therapy was associated with systemic doxycycline 100 mg/day, for two weeks after an initial dose of 200 mg, started on the day before the first scaling and root planning session. Patients of the PD group had no access to information about antibiotics administration to patients of the PD+DM group.
  Other Names: Doxilegrand, Legrand, São Bernardo do Campo, SP, Brazil.
  Arms: Chronic periodontitis + type 2 diabetes
Procedure: Non-surgical periodontal therapy — A program of plaque control with dental prophylaxis and oral hygiene instruction, and the scaling and root planning sessions were included in the non-surgical periodontal therapy. The scaling and root planning was performed by the same operator using curettes and an ultrasonic device, and it was inspected for a second operator. Oral hygiene was reviewed after a week and after a month of periodontal disinfection, followed by dental prophylaxis.
  Other Names: Scaling and root planning
  Arms: chronic periodontitis

SUMMARY:
The purpose of the study was to monitor the activity of periodontal disease and suggest potential biomarkers related to active periodontal disease in patients with chronic periodontitis (PD) associated or not with type 2 diabetes mellitus (DM), based on the evaluation of the profile of gene expression of periodontal sites and the evaluation of inflammatory salivary proteins. Two hundred and five periodontal patients were enrolled, but only 41 exhibited ≥ 1 mm attachment loss in at least three periodontal site (active sites) 2 months after non-surgical periodontal therapy. The final sample was: 21 patients with chronic periodontitis (PD group) and 20 with chronic periodontitis and diabetes (PD+DM group). Fifteen periodontal- and systemically healthy patients were included as control group. Saliva collection, glycated hemoglobin measurement, periodontal examination and radiographs were conducted before and 2 months after non-surgical periodontal therapy. Radiographic subtraction was performed from pairs of the radiographs. Measurements of the areas with density loss were recorded. Gingival biopsies of active and non-active sites with similar clinical parameters were harvested for Real Time Polymerase Chain Reaction Array gene expression analysis. Saliva samples were analyzed by Multiplex Cytokine Profiling Immunoassay for analysis of protein expression. The clinical attachment loss mean was higher in the PD+DM group (p<0.05). There was a high correlation between clinical attachment loss and darkened radiographic areas in active sites of the PD group and PD+DM group. When compared PD group to PD+DM, patients with diabetes had an up-regulated profile. Active sites of the PD group showed nine genes (specific chemokines, interleukins and receptors) differentially expressed with an up-regulated profile. Active sites of the PD+DM group showed six genes (specific chemokines, interleukins and receptors) differentially expressed with an up-regulated profile. After periodontal therapy, there was a reduction of some salivary proteins in both periodontal groups, but not significant. In conclusion, it was possible to identify genes differentially expressed in active sites from both groups, which may be considered useful in indicating potential biomarkers for the diagnosis of periodontitis; salivary proteins show a trend in distinguishing the standard of health and disease and may be used in the future as potential biomarkers of periodontitis with or without diabetes.

DETAILED DESCRIPTION:
This case-control longitudinal study was carried out at University of São Paulo between March 2009 and June 2012 as a joint collaboration of the Department of Oral Surgery and Periodontology and the Department of Internal Medicine, Division of Endocrinology and Metabolism. It was reviewed and approved by the Institutional Human Ethics Research Committee of the Ribeirão School of Dentistry - University of Sao Paulo (process n. 2009.1.88.58.7).

The clinical attachment loss above 1 mm was determined according to the tolerance method adapted to the computerized periodontal probe, considering the standard deviation of 0.3 mm for the electronic probe multiplied by 3. Teeth with prosthesis or furcation lesions were not considered. The periodontal sites that had this clinical attachment were called active sites.

Before beginning the initial clinical examination, a supragingival scaling with ultrasonic device was performed to facilitate the examination. The clinical parameters evaluated were: probing pocket depth, relative clinical attachment level and bleeding on probing were recorded at six sites per tooth with the aid of a computerized periodontal probe. To reduce the variations between baseline and 12-month evaluations, an acrylic stent was used to standardize the position of the computerized periodontal probe. Bleeding on probing was assessed according to presence or absence of bleeding up to 20 seconds after probing. The plaque index, presence or absence of biofilm, was recorded at four sites per tooth. It was also verified the furcation involvement with the aid of a manual periodontal probe.

All clinical parameters were recorded two weeks after supragingival scaling (baseline) and two months after non-surgical periodontal therapy by one-blinded calibrated examiner. A calibration exercise was performed to achieve acceptable intraexaminer reproducibility.

For the metabolic control assessment, the HbA1c levels were analyzed in patients from both groups at baseline and two months after non-surgical periodontal therapy, at the Endocrinology Clinic of the Ribeirão Preto School of Medicine, University of São Paulo. All diabetics were under the supervision of an endocrinologist advised to communicate any change in medicine intake or diet.

A program of plaque control with dental prophylaxis and oral hygiene instruction, and the scaling and root planning sessions were performed by the same operator using curettes and an ultrasonic device in PD and PD+DM groups. All scaling and root planning procedures were inspected for a second operator. Oral hygiene was reviewed after a week and after a month of periodontal disinfection, followed by dental prophylaxis.

In PD+DM group, the non-surgical periodontal therapy was associated with systemic doxycycline 100 mg/day, for two weeks after an initial dose of 200 mg, started on the day before periodontal therapy. Patients of the PD group had no access to information about antibiotics administration to patients of the PD+DM group.

Non-stimulated whole expectorated saliva was collected (~ 3 ml) from each subject into sterile tubes. Subjects were refrained from eating, drinking, and oral hygiene for 2 hours prior to saliva collection. Saliva samples were placed on ice immediately and aliquoted prior to freezing at -80º Celsius. Samples were thawed and analyzed within 6 months of collection.

A complete series of radiographs was taken in each patient at baseline, using the paralleling technique. Two months after periodontal therapy, radiographs were taken with the same technique in teeth with active periodontal sites. Thereafter, the radiographs were digitized in tagged image file format (TIFF) on a scanner. Digital subtraction radiographs were performed with the baseline and 2-month radiographs using specific software. Only teeth with interproximal sites with periodontal disease activity were included in this analysis. Changes between radiographs were depicted as a darkened area for loss of alveolar bone mass. These areas were measured (mm2) using specific measurements software. As in the clinical examination, it was performed intra-examiner calibration for the measurements of areas of radiographic density loss.

Gingival tissue samples were obtained from active sites of the each patient in both groups during regular periodontal surgery. The excised gingival collar was then carefully removed from the roots and the alveolar process. Gingival biopsy comprised epithelial and connective tissues. The samples are immediately submerged into liquid nitrogen to be then stored at -80º Celsius for RNA extraction and gene expression analysis.

Total RNA from biopsies was extracted using the Trizol reagent according to the directions supplied by the manufacturer. From 1 µg of total RNA, a strand of complementary DNA (cDNA) was synthesized through a reverse transcription reaction according to the directions supplied by the manufacturer. At the end of this reaction, cDNA was stored at -20º Celsius for later use. The Real Time Polymerase Chain Reaction (PCR) Array allowed simultaneous analysis of 84 genes involved in specific signaling pathways. The genes included in PCR array plates for human inflammatory cytokines and receptors.

ELIGIBILITY:
Inclusion Criteria:

* adults aged between 35 to 65 years old;
* a minimum of 14 natural teeth, 10 of which should be posterior teeth;
* periodontitis case definition was the presence of five teeth with a probing pocket depth of ≥ 5 mm and clinical attachment loss of ≥ 3 mm;
* type 2 diabetes for at least 5 years and with glycated hemoglobin level > 7%.

Exclusion Criteria:

* smoking within the last 5 years;
* pregnancy or lactating;
* use of antibiotics or periodontal therapy in the previous six months;
* concomitant medical therapy, except for diabetic condition;
* other inflammatory conditions;
* major diabetic complications such as retinopathy, nephropathy, neuropathy and atherosclerosis.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2009-03; Primary Completion 2011-09 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
clinical attachment level | baseline and two months
  relative clinical attachment level (rCAL) was recorded at six sites per tooth with the aid of a computerized periodontal probe.

SECONDARY OUTCOMES:
Gene expression | Two months
  Gingival tissue samples were obtained from periodontal sites (active or non-active) of the each patient in both groups during regular periodontal surgery. The samples are immediately submerged into liquid nitrogen to be then stored at -80º Celsius for RNA extraction and cDNA synthesis. The Real Time-PCR Array allowed simultaneous analysis of 84 genes involved in specific signaling pathways, including specific human inflammatory cytokines and receptors.
Salivary proteins levels | baseline and two months
  Non-stimulated whole expectorated saliva was collected (~ 3 ml) from each subject into sterile tubes and stored at -80º Celsius. The salivary inflammatory proteins levels were identified simultaneously using Multiplex Cytokine Profiling Assay, which allows the simultaneous detection of multiple analytes in saliva sample size.

OTHER OUTCOMES:
Probing pocket depth | baseline and two months
  It was recorded at six sites per tooth with the aid of a computerized periodontal probe.
Bleeding on probing | baseline and two months
  It was recorded at six sites per tooth with the aid of a computerized periodontal probe, and it was assessed according to presence or absence of bleeding up to 20 seconds after probing.
Plaque index | baseline and two months
  It was recorded at four sites per tooth to assess presence or absence of dental biofilm.
Glycated hemoglobin level | baseline and two months
  Metabolic control assessment
Density loss | baseline and two months
  A complete series of radiographs was taken in each patient at baseline, using the paralleling technique. Two months after periodontal therapy, radiographs were taken with the same technique in teeth with active periodontal sites. The radiographs were digitized in tagged image file format (TIFF) on a scanner. Digital subtraction radiographs were performed with the baseline and 2-month radiographs using specific software. Changes between radiographs were depicted as a darkened area for loss of alveolar bone mass. These areas were measured (mm2) using specific measurements software.

CONTACTS AND LOCATIONS:
Overall Officials: Priscila P Costa, PhD, Principal Investigator — Department of Oral Surgery and Periodontology - Ribeirão Preto School of Dentistry, University of São Paulo
Locations (1):
- Mario Taba Jr, Ribeirão Preto, São Paulo, Brazil